CLINICAL TRIAL: NCT06295159
Title: Neoadjuvant and Adjuvant Anti-PD1 or Combinations for Locoregionally Advanced Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-22574
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Melanoma Stage III; Melanoma Stage IV; Advanced Melanoma; Melanoma
Keywords: Melanoma; Anti-PD1; Locoregionally Advanced Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; relatlimab; Opdualag; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part 1, Arm A: Nivolumab (Experimental): PD-L1 positive patients will be given Nivolumab 480 mg I.V. over 30 minutes (-/+ 10 minutes) every 4 weeks (every cycle) for 2 a total of 2 cycles.
  Interventions: Drug: Nivolumab
- Part 1, Arm B: Nivolumab- Relatlimab-rmbw (Experimental): PD-L1 negative patients will be given a combination of Nivolumab 480 mg with Relatlimab 160 mg I.V. over 60 minutes (-/+ 10 minutes) every 4 weeks (every cycle) for a total of 2 cycles.
  Interventions: Drug: Nivolumab + Relatlimab
- Part 1, Arm C: Nivolumab plus ipilimumab (Experimental): PD-L1 negative patients will be given 3 mg/kg of Nivolumab plus 1 mg/kg of Ipilimumab I.V. each given over 30 minutes (-/+ 10 minutes) every 4 weeks (every cycle) for a total of 2 cycles.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Part 2, Arm A: Ipilimumab + Nivolumab-Relatimab-rmbw (Experimental): Systemic therapy naïve locoregionally advanced melanoma patients will be given the fixed dose combination of 480 mg of nivolumab with 160 mg of relatlimab I.V. over 60 minutes (-/+ 10 minutes) every 4 weeks (every cycle) for a total of 2 cycles.
  In addition, a single dose of 1 mg/kg ipilimumab I.V. will be given on C1D1.
  Interventions: Drug: Nivolumab + Relatlimab; Drug: Ipilimumab
- Part 2, Arm B1: Triplet Combination Therapy Ipilmumab + Nivolumab-Relatlimab-rmbw (Experimental): Patients with locoregionally advanced melanoma that is refractory to systemic adjuvant therapy will be given the fixed dose combination of 480 mg of nivolumab with 160 mg or relatlimab I.V. over 60 minutes (-/+ 10 minutes) every 4 weeks (every cycle) for a total of 2 cycles.
  In addition, a single dose of 1 mg/kg ipilimumab I.V. will be given on C1D1.
  Interventions: Drug: Nivolumab + Relatlimab; Drug: Ipilimumab
- Part 2, Arm B2: Doublet Combination Therapy Nivolumab-Relatlimab-rmbw (Experimental): Patients with locoregionally advanced melanoma that is refractory to systemic adjuvant therapy will be given the fixed dose combination of 480 mg of nivolumab with 160 mg of relatlimab I.V. over 60 minutes (-/+ 10 minutes) every 4 weeks (every cycle) for a total of 2 cycles.
  Interventions: Drug: Nivolumab + Relatlimab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a fully human immunoglobulin (Ig) G4 monoclonal antibody directed against the negative immunoregulatory human cell surface receptor programmed death-1 (PD-1, PCD-1) with immune checkpoint inhibitory and antineoplastic activities. Upon administration, nivolumab binds to and blocks the activation of PD-1, an immunoglobulin superfamily (IgSF) transmembrane protein, by its ligands programmed cell death ligand 1 (PD-L1), which is overexpressed on certain cancer cells, and programmed cell death ligand 2 (PD-L2), which is primarily expressed on antigen-presenting cells (APCs). This results in the activation of T cells and cell-mediated immune responses against tumor cells. Activated PD-1 negatively regulates T-cell activation and plays a key role in tumor evasion from host immunity.
  Other Names: Opdivo
  Arms: Part 1, Arm A: Nivolumab; Part 1, Arm C: Nivolumab plus ipilimumab
Drug: Nivolumab + Relatlimab — Opdualag (Nivolumab and Relatlimab-rmbw) is a combination formulation composed of nivolumab, a human immunoglobulin (Ig) G4 monoclonal antibody directed against the negative immunoregulatory human cell surface receptor programmed death-1 (PD-1, PCD-1), and relatlimab-rmbw, a human IgG4 monoclonal antibody directed against the inhibitor receptor lymphocyte activation gene-3 (LAG-3). Nivolumab binds to and blocks the activation of PD-1 by its ligands programmed cell death ligand 1 (PD-L1), which is overexpressed on certain cancer cells, and programmed cell death ligand 2 (PD-L2), which is primarily expressed on antigen-presenting cells (APCs). This prevents PD-1-mediated signaling and PD-1-mediated inhibition of the immune response. Relatlimab binds to LAG-3 on tumor infiltrating lymphocytes (TILs) and prevents LAG-3 binding to major histocompatibility complex (MHC) class II. This prevents LAG-3-mediated signaling and LAG-3-mediated inhibition of the immune response.
  Other Names: Opdualag
  Arms: Part 1, Arm B: Nivolumab- Relatlimab-rmbw; Part 2, Arm A: Ipilimumab + Nivolumab-Relatimab-rmbw; Part 2, Arm B1: Triplet Combination Therapy Ipilmumab + Nivolumab-Relatlimab-rmbw; Part 2, Arm B2: Doublet Combination Therapy Nivolumab-Relatlimab-rmbw
Drug: Ipilimumab — Ipilimumab is a type of monoclonal antibody and a type of immune checkpoint inhibitor that may block CTLA-4 and help the immune system kill cancer cells. Ipilimumab binds to the protein CTLA-4 to help immune cells kill cancer cells better and is used to treat many different types of cancer. These include cancers that have certain mutations (changes) in genes involved in DNA repair.
  Other Names: Yervoy
  Arms: Part 1, Arm C: Nivolumab plus ipilimumab; Part 2, Arm A: Ipilimumab + Nivolumab-Relatimab-rmbw; Part 2, Arm B1: Triplet Combination Therapy Ipilmumab + Nivolumab-Relatlimab-rmbw

SUMMARY:
The purpose of this study is to determine if neoadjuvant (treatment before surgery) immunotherapy treatment based on tumor biomarkers results in better participant outcomes. Immunotherapy is the treatment of disease by using a person's own immune system.

This study is divided into 2 sub-studies/parts designated Part 1 and Part 2 that will enroll in sequence starting with Part 1 followed by Part 2.

ELIGIBILITY:
Inclusion Criteria:

* This study is divided into 2 sub-studies/parts designated Part 1 and Part 2 that will enroll in sequence starting with Part 1 followed by Part 2. In Part 2, Part 2 Cohort A and Part 2 Cohort B will enroll simultaneously. Inclusion criteria apply to Part 1 and Part 2 unless otherwise specified.
* Voluntarily agree to participate by giving signed, dated, and written informed consent prior to any study-specific procedures.
* 18 years of age or older
* Histologic diagnosis of melanoma (cutaneous, acral, mucosal or unknown primary) belonging to the following American Joint Committee on Cancer (AJCC) 8th edition TNM stages (Tx or T1-4) and (N1b, N1c, N2b, N2c, N3b or N3c) and/or (M1a).
* Requirements for prior systemic therapy for melanoma are as follows:

  1. Sub-study Part 1: No prior systemic therapy for melanoma (N=30).
  2. Sub-study Part 2 Cohort A: No prior systemic therapy for melanoma (N=20)
  3. Sub-study Part 2 Cohort B: Locoregionally advanced melanoma that is refractory to systemic adjuvant therapy (anti-PD1-based or BRAF-MEK inhibitors) (N=40).

This excludes patients who previously received adjuvant or neoadjuvant anti-PD1 plus anti-LAG3 or anti-PD1 plus anti-CTLA4.

Participants who experienced progression or recurrence after anti-PD1 as monotherapy or other combinations or after BRAF-MEK inhibition would be eligible.

Participants who have previously experienced prior high-grade (grade 3 or 4 by CTCAE criteria) immune related adverse events with immune checkpoint inhibitors are not eligible.

* Must be considered surgically operable and may present as any of the following groups:

  1. Primary melanoma with clinically apparent regional lymph node metastases, confirmed by pathological diagnosis.
  2. Clinically detected recurrence of melanoma at regional lymph node basin(s), confirmed by pathological diagnosis.
  3. Clinically or histologically detected primary melanoma involving multiple regional nodal groups, confirmed by pathological diagnosis.
  4. Clinically detected single site of nodal metastatic melanoma arising from an unknown primary, confirmed by pathological diagnosis.
  5. Participants with in-transit or satellite metastases with or without lymph node involvement are allowed if they are considered surgically resectable at Screening by the treating surgical oncologist.
  6. Participants with distant cutaneous/subcutaneous, soft tissue or nodal metastases with or without regional lymph node involvement are allowed if they are considered potentially surgically resectable and can be biopsied at Screening by the treating surgical oncologist. Elevated LDH is not an exclusion.
  7. Elevated LDH is not an exclusion.
* Participants are eligible for this study either at presentation for primary melanoma with concurrent regional nodal and/or in-transit or distant metastasis, or at the time of clinically detected nodal, in transit, or distant recurrence.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function within 28 days of Cycle 1 Day 1 (C1D1)
* Participants must provide a sufficient and adequate formalin-fixed paraffin-embedded (FFPE) tumor tissue sample from the most recent biopsy of a tumor lesion, obtained within 90 days from signing informed consent form (ICF). If recent tumor tissue is unavailable or inadequate, a fresh biopsy will be required, unless the principal investigator agrees that it is not safe/feasible.
* Participants must be evaluated by standard-of-care full body imaging studies, the choice of which is decided by the treating physician investigator.
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test at screening (within 72 hours of first dose of study medication) in accordance with the standard of care for WOCBP.
* WOCBP must agree to use highly effective contraceptive measures starting with the screening visit through 5 months after the last dose of study treatment. Highly effective contraception is as stipulated in national or local guidelines.
* Male participants with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the study starting with the screening visit through 5 months after the last dose of study treatment is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.
* Willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

* Pregnancy or lactation.
* Treatment with another investigational drug or other systemic intervention for melanoma within 4 weeks of initiation of study drugs. Patients must not have radiotherapy within the preceding 2 weeks. Patients must have recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants must be at least 4 weeks from major surgery and have fully recovered from any effects of surgery and be free of significant detectable infection.
* Ocular or uveal melanoma.
* Bowel obstruction or impending bowel obstruction within the past 3 months.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure or serious uncontrolled cardiac arrhythmia requiring medication.
* Active or history of brain metastases or leptomeningeal metastases.
* Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to the first dose of study treatment, i.e., patients with a history of prior malignancy are eligible if treatment was completed at least 2 years before the first dose of study treatment and the patient has no evidence of disease. Participants with history of prior early-stage basal/squamous cell skin cancer, low-risk prostate cancer eligible for active surveillance or noninvasive or in situ cancers who have undergone definitive treatment at any time are also eligible.
* Treatment with one of the following classes of drugs within the delineated time window prior to C1D1:

  1. Cytotoxic, targeted therapy or other investigational therapy within 3 weeks.
  2. mAbs, antibody-drug conjugates, radioimmunoconjugates, or similar therapy, within 4 weeks, or 5 half-lives, whichever is shorter.
  3. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccine or booster < 7 days before C1D1. For vaccines requiring more than 1 dose, the full series should be completed prior to C1D1, when feasible. Booster shot not required but also must be administered > 7 days from C1D1 or > 7 days from future cycle on study.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Any evidence of current interstitial lung disease (ILD) or pneumonitis or a prior history of ILD or non-infectious pneumonitis requiring high-dose glucocorticoids.
* History of allogeneic organ transplant.
* Psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) within 14 days or another immunosuppressive medication within 30 days of the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years before starting treatment, i.e., with use of disease-modifying agents or immunosuppressive drugs.
* History or current evidence of any condition, co-morbidity, therapy, any active infections, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* Pregnant or breastfeeding or WOCBP who are not willing to employ effective birth control from screening to 5 months after the last dose of study treatment (whichever is later).
* Previous SARS-CoV-2 infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to C1D1.
* Uncontrolled infection with human Immunodeficiency virus (HIV). Patients on stable highly active antiretroviral therapy (HAART) with undetectable viral load and normal CD4 counts for at least 6 months prior to study entry are eligible. Serological testing for HIV at screening is not required.
* Known to be positive for hepatitis B virus (HBV) surface antigen, or any other positive test for HBV indicating acute or chronic infection. Patients who are receiving or who have received anti-HBV therapy and have undetectable HBV DNA for at least 6 months prior to study entry are eligible. Serological testing for HBV at screening is not required. Known active co-infection with hepatitis B and hepatitis C or with hepatitis B and hepatitis D is an exclusion.
* Known active hepatitis C virus (HCV) as determined by positive serology and confirmed by polymerase chain reaction (PCR). Patients on or who have received antiretroviral therapy are eligible provided they are virus-free by PCR for at least 6 months prior to study entry. Serological testing for HCV at screening is not required.
* Dependence on total parenteral nutrition.
* Troponin T (TnT) or I (TnI) > 2× institutional ULN. Participants with TnT or TnI levels between > 1 to 2 × ULN will be permitted if repeat levels within 24 hours are ≤ 1 × ULN. If TnT or TnI levels are between >1 to 2 × ULN within 24 hours, the participant must undergo a cardiology consultation and cardiac evaluation and be considered for treatment, based on a favorable benefit/risk assessment by the Investigator. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 × ULN, the participant must undergo a cardiology consultation and cardiac evaluation and be considered for treatment, based on a favorable benefit-risk assessment by the Investigator.
* Left ventricular ejection fraction (LVEF) assessment with documented LVEF < 50% by either transthoracic echocardiogram (TTE) or multigated acquisition (MUGA) scan (TTE preferred test) within 6 months prior to start of study treatment.
* Participants with a history of myocarditis and/or current diagnosis of myocarditis, regardless of etiology.
* Participants must not have a history of allergy or hypersensitivity to study intervention components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Pathologic Major Response (pMR) | Up to 36 Months
  The pathologic response rate will be measured by evaluation of the residual viable tumor (RVT).
  Pathologic Major Response (pMR) is defined as near complete response (pCR) measured as ≤10% RVT + complete response (pCR) measured as 0% RVT.

SECONDARY OUTCOMES:
Preoperative Radiologic Response Rate | Up to 8 Weeks
  The Preoperative Radiologic Response Rate will be measured utilizing RECIST v.1.1.
Complete Pathologic Response Rate (pCR) | Up to 36 Months
  The pathologic response rate will be measured by evaluation of the residual viable tumor (RVT).
  Pathologic Complete Response (pCR) is defined as 0% RVT.
Partial Pathologic Response Rate (pPR) | Up to 36 Months
  The pathologic response rate will be measured by evaluation of the residual viable tumor (RVT).
  Pathologic Partial Response (pPR) is defined as 10-50% RVT.
Non-Response Pathologic Response Rate (pNR) | Up to 36 Months
  The pathologic response rate will be measured by evaluation of the residual viable tumor (RVT).
  Pathologic Non-Response (pNR) is defined as 50-100% RVT.
Progression Free Survival (PFS) | Up to 36 Months
  Progression Free Survival (PFS) will be measured from the date of start of treatment to the investigator-determined date of progression or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 36 Months
  Overall Survival (OS) will be measured from the initial date of study registration/randomization to the recorded date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org/clinical-trials-research/clinical-trials/